CLINICAL TRIAL: NCT05654519
Title: Comparison of Pericapsular Nerve Group Block with Lateral Femoral Cutaneous Nerve Block and Quadratus Lumborum Block for Total Hip Arthroplasty
Brief Title: Comparison of Pericapsular Nerve Group Block and Quadratus Lumborum Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Necmettin Erbakan Üniversitesi (Other)
Responsible Party: Principal Investigator, Alper Kilicaslan, Clinical Professor, Konya Necmettin Erbakan Üniversitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-541
Record Dates: First submitted 2022-11-30; First posted 2022-12-16 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2023-04

CONDITIONS: Total Hip Surgery; Pericapsular Nerve; Quadratus Lumborum
Keywords: Total Hip Surgery; PENG block; QLB

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient, and the outcomes assessor who performs postoperative pain evaluation will not know the group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group QL Block (Active Comparator): A convex transducer will be placed in the transverse plane on the flank cranial to the iliac crest to visualise the transverse process of the 4th lumbar vertebra, erector spina, quadratus lumborum and psoas muscles as a 'Shamrock sign'. The needle will inserted in to the fascial plane between the quadratus lumborum and psoas muscles and 30 ml bupivacaine 0.25% will be administered.
  Interventions: Drug: PENG/LFCN and QL Blocks
- Group PENG+LFCN Block (Active Comparator): A linear probe will be placed on the anterior inferior iliac crest in the transverse plane while the patient is in the supine position. After rotating 45 degrees, the pubic ramus, femoral artery and psoas muscle will be visualized. Puncture will be performed in a lateromedial direction until the needle tip reached the plane between the iliopsoas tendon and the iliopubic eminence After a negative aspiration test, 25 ml bupivacaine 0.25% will be injected.
  Then, the lateral femoral cutaneous nerve (LFCN) block was performed using linear US probe (10-18 MHz).The LFCN will be localized, infero-medially to the antero-superior iliac spine, laterally to the sartorius muscle and 5 ml of bupivacaine 0.25% will be carefully injected.
  Interventions: Drug: PENG/LFCN and QL Blocks

INTERVENTIONS:
Drug: PENG/LFCN and QL Blocks — Bupivacaine 0.25% injection

SUMMARY:
Adequate pain management following total hip arthroplasty (THA) is a key component for patient satisfaction and early ambulation. However, due to the complexity of the innervation of the hip joint, the most appropriate anaesthetic and analgesic technique for THA remains unclear. A femoral nerve block is commonly performed and well established but is associated with motor weakness. Recently, the pericapsular nerve group (PENG) block has been introduced as an effective choice which targets the articular branches of the hip. The quadratus lumborum block (QLB) is a relatively new regional block that has been reported to provide effective analgesia for THA.

The main objective of this study is to compare the effectiveness of the ultrasound-guided PENG block technique compared to QLB block in terms of efficacy of pain control and the safety profile after total hip arthroplasty under spinal anesthesia.

DETAILED DESCRIPTION:
The patients will be randomly classified into two equal groups (40 patients each). Group allocation will be done by computer generated random numbers and closed opaque sealed envelopes. The study will be designed to be double blind as all patients and outcomes assessor will be blinded to group assignment.

Patients will be randomized to one of three equal groups:

Group I (n= 40 patients): Patients in this group will receive an ipsilateral single shot of QLB (30 ml of plain bupivacaine 0.25%) after surgery using ultrasonographic guidance.

Group II(n= 40 patients): patients in this group will receive an ipsilateral single-shot of PENG block (25 ml of plain bupivacaine 0.25%) and LFCN block (5 ml of plain bupivacaine 0.25%) after surgery using ultrasonographic guidance.

ELIGIBILITY:
Inclusion Criteria:

Physical status according to American Society of Anesthesiologists (ASA ) I-III

Exclusion Criteria:

* Younger than 40 years old and older than 85
* Patients undergoing general anesthesia
* Allergy or intolerance to one of the study medications
* Infection of the skin at the site of the needle puncture,
* Patients who do not accept the procedure
* History of bleeding diathesis
* ASA IV,
* Chronic gabapentin/pregabalin,opioid use
* Hepatic or renal insufficiency
* Previous operation on the same hip
* BMI >40

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
Pain scores | Changes from baseline opioid consumption at postoperative 0, 2, 6, 12 and 24 hours
  Numerical Rating Scale-NRS (0 = no pain and 10 = worst imaginable painranged from 0 to 10)
Opioid consumption | Changes from baseline opioid consumption at postoperative 0, 2, 6, 12 and 24 hours
  Mean opioid consumption in morphine equivalents

SECONDARY OUTCOMES:
Quadriceps muscle strength | Postoperative 24 hours period
  Quadriceps motor function will be tested with the patient supine and with the hip and knee flexed at 45º and 90º, respectively
Presence of postoperative nausea, vomiting, pruritus, urinary retention, respiratory depression | Postoperative 24 hours period
  Presence of postoperative nausea, vomiting, pruritus, urinary retention, respiratory depressio
Patient satisfaction | Postoperative 24 hours period
  Patients asked whether they would choose the same anaesthetic management in a future operation: Yes/No

CONTACTS AND LOCATIONS:
Locations (1):
- Alper KILICASLAN, Konya, Turkey (Türkiye)

REFERENCES:
- [Background] Hussain N, Brull R, Speer J, Hu LQ, Sawyer T, McCartney CJL, Abdallah FW. Analgesic benefits of the quadratus lumborum block in total hip arthroplasty: a systematic review and meta-analysis. Anaesthesia. 2022 Oct;77(10):1152-1162. doi: 10.1111/anae.15823. Epub 2022 Aug 10. PMID 35947882
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657